CLINICAL TRIAL: NCT01443637
Title: COronary CT Angiography Evaluation For Clinical Outcomes: An International Multicenter Registry
Brief Title: COroNary CT Angiography Evaluation For Clinical Outcomes: An InteRnational Multicenter Registry (CONFIRM)
Acronym: CONFIRM
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1310014468
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Cardiovascular Disease
Keywords: Coronary Artery Disease; CAD; Atherosclerosis; Myocardial Infarction; MI; CONFIRM; Coronary Computed Tomographic Angiography; CCTA
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary CT Angiography (CCTA): Patients included in the CONFIRM Registry are those that have previously undergone clinically-indicated CCTA as part of their standard of care.

SUMMARY:
The CONFIRM study was developed to examine the prognostic value of cardiac computed tomographic angiography (CCTA) findings for prediction of future adverse cardiac events related to coronary artery disease (CAD) in a large, international patient population. The purpose of this multicenter registry is to correlate coronary and non-coronary cardiac findings by CCTA with demographic and clinical data for refinement of risk stratification of individuals with suspected or known CAD.

DETAILED DESCRIPTION:
Coronary computed tomographic angiography (CCTA) of 64-detector rows or greater represents a novel noninvasive anatomic method for evaluation of patients with suspected coronary artery disease (CAD). Early studies suggest a potential for prognostic risk assessment by CCTA findings but were limited by small patient cohorts or single centers. The CONFIRM Registry is a large, prospective, multinational dynamic observational study of patients undergoing CCTA. The primary aim of CONFIRM is to determine the prognostic value of CCTA findings for the prediction of future adverse CAD events.

The CONFIRM registry currently represents 27,125 consecutive patients at 12 cluster sites in 6 countries in North America, Europe, and Asia. CONFIRM sites were chosen on the basis of adequate CCTA volume, site CCTA proficiency, and local demographic characteristics and medical facilities to ensure a broad-based sample of patients. Patients comprising the present CONFIRM cohort include those with suspected but without known CAD, with known CAD, or asymptomatic persons undergoing CAD evaluation. A data dictionary comprising a wide array of demographic, clinical, and CCTA findings was developed by the CONFIRM investigators and is uniformly used for all patients. Patients are followed up after CCTA performance to identify adverse CAD events, including death, myocardial infarction, unstable angina, target vessel revascularization, and CAD-related hospitalization.

ELIGIBILITY:
All consecutive patients at cluster sites meeting all inclusion criteria undergoing CCTA of 64-detector rows or greater will be included within the CONFIRM registry.

Inclusion Criteria:

1. Age > 18 years
2. Evaluation by CCTA with 64-detector rows or greater for CAD evaluation as part of standard of care
3. Interpretable CCTA
4. Prospective data collection for CAD risk factors.

Exclusion Criteria:

No explicit patient exclusion criteria are defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of patients at multiple international centers undergoing clinically-indicated coronary CT angiography as part of their standard of care.
Sampling Method: Probability Sample
Enrollment: 34000 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Coronary and non-coronary cardiac findings by CCTA | yearly
  Identify, quantify, and integrate coronary and noncoronary cardiac findings by Coronary computed tomographic angiography (CCTA) with demographic and clinical data for refinement of risk stratification of persons with suspected or known CAD.

CONTACTS AND LOCATIONS:
Overall Officials: Leslee J Shaw, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (20):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cardiovascular Medical Group of Southern California, Los Angeles, California
  - Harbor UCLA, Los Angeles, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Capital Cardiology Associates, Albany, New York
  - Weill Cornell Medical Center, New York, New York
  - Tenessee Heart and Vascular Institute, Hendersonville, Tennessee
- Medical University Innsbruck, Innsbruck, Austria
- Canada (2):
  - Providence Health Care, Vancouver, British Columbia
  - Ottawa Heart Institute, Ottawa, Ontario
- Germany (2):
  - University of Giessen, Giessen
  - Deutsches Herzzentrum Munchen, Munich
- University of Parma, Parma, Italy
- South Korea (2):
  - Seoul National University College of Medicine, Seoul
  - Severance Cardiovascular Hospital, Seoul
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Min JK, Dunning A, Lin FY, Achenbach S, Al-Mallah MH, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng V, Chinnaiyan KM, Chow B, Delago A, Hadamitzky M, Hausleiter J, Karlsberg RP, Kaufmann P, Maffei E, Nasir K, Pencina MJ, Raff GL, Shaw LJ, Villines TC. Rationale and design of the CONFIRM (COronary CT Angiography EvaluatioN For Clinical Outcomes: An InteRnational Multicenter) Registry. J Cardiovasc Comput Tomogr. 2011 Mar-Apr;5(2):84-92. doi: 10.1016/j.jcct.2011.01.007. Epub 2011 Feb 1. PMID 21477786
- [Background] Cho I, Al'Aref SJ, Berger A, O Hartaigh B, Gransar H, Valenti V, Lin FY, Achenbach S, Berman DS, Budoff MJ, Callister TQ, Al-Mallah MH, Cademartiri F, Chinnaiyan K, Chow BJW, DeLago A, Villines TC, Hadamitzky M, Hausleiter J, Leipsic J, Shaw LJ, Kaufmann PA, Feuchtner G, Kim YJ, Maffei E, Raff G, Pontone G, Andreini D, Marques H, Rubinshtein R, Chang HJ, Min JK. Prognostic value of coronary computed tomographic angiography findings in asymptomatic individuals: a 6-year follow-up from the prospective multicentre international CONFIRM study. Eur Heart J. 2018 Mar 14;39(11):934-941. doi: 10.1093/eurheartj/ehx774. PMID 29365193
- [Background] Lee JH, Han D, Hartaigh BO, Gransar H, Lu Y, Rizvi A, Park MW, Roudsari HM, Stuijfzand WJ, Berman DS, Callister TQ, DeLago A, Hadamitzky M, Hausleiter J, Al-Mallah MH, Budoff MJ, Kaufmann PA, Raff G, Chinnaiyan K, Cademartiri F, Maffei E, Villines TC, Kim YJ, Leipsic J, Feuchtner G, Pontone G, Andreini D, Marques H, Rubinshtein R, Achenbach S, Shaw LJ, Chang HJ, Bax J, Chow B, Cury RC, Gomez M, Jones EC, Lin FY, Min JK, Pena JM. Influence of symptom typicality for predicting MACE in patients without obstructive coronary artery disease: From the CONFIRM Registry (Coronary Computed Tomography Angiography Evaluation for Clinical Outcomes: An International Multicenter Registry). Clin Cardiol. 2018 May;41(5):586-593. doi: 10.1002/clc.22940. Epub 2018 May 11. PMID 29521447
- [Background] van Rosendael AR, Maliakal G, Kolli KK, Beecy A, Al'Aref SJ, Dwivedi A, Singh G, Panday M, Kumar A, Ma X, Achenbach S, Al-Mallah MH, Andreini D, Bax JJ, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJW, Cury RC, DeLago A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann PA, Kim YJ, Leipsic JA, Maffei E, Marques H, Pontone G, Raff GL, Rubinshtein R, Shaw LJ, Villines TC, Gransar H, Lu Y, Jones EC, Pena JM, Lin FY, Min JK. Maximization of the usage of coronary CTA derived plaque information using a machine learning based algorithm to improve risk stratification; insights from the CONFIRM registry. J Cardiovasc Comput Tomogr. 2018 May-Jun;12(3):204-209. doi: 10.1016/j.jcct.2018.04.011. Epub 2018 Apr 30. PMID 29753765
- [Background] Cho YK, Nam CW, Koo BK, Schulman-Marcus J, Hartaigh BO, Gransar H, Lu Y, Achenbach S, Al-Mallah M, Andreini D, Bax JJ, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJW, Cury RC, Delago A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann PA, Kim YJ, Leipsic J, Maffei E, Marques H, Pontone G, Raff GL, Rubinshtein R, Shaw LJ, Villines TC, Berman DS, Jones EC, Pena JM, Lin FY, Min JK. Usefulness of baseline statin therapy in non-obstructive coronary artery disease by coronary computed tomographic angiography: From the CONFIRM (COronary CT Angiography EvaluatioN For Clinical Outcomes: An InteRnational Multicenter) study. PLoS One. 2018 Dec 12;13(12):e0207194. doi: 10.1371/journal.pone.0207194. eCollection 2018. PMID 30540755
- [Background] Lee JH, Rizvi A, Hartaigh BO, Han D, Park MW, Roudsari HM, Stuijfzand WJ, Gransar H, Lu Y, Callister TQ, Berman DS, DeLago A, Hadamitzky M, Hausleiter J, Al-Mallah MH, Budoff MJ, Kaufmann PA, Raff GL, Chinnaiyan K, Cademartiri F, Maffei E, Villines TC, Kim YJ, Leipsic J, Feuchtner G, Pontone G, Andreini D, Marques H, de Araujo Goncalves P, Rubinshtein R, Achenbach S, Shaw LJ, Chow BJW, Cury RC, Bax JJ, Chang HJ, Jones EC, Lin FY, Min JK, Pena JM. The Predictive Value of Coronary Artery Calcium Scoring for Major Adverse Cardiac Events According to Renal Function (from the Coronary Computed Tomography Angiography Evaluation for Clinical Outcomes: An International Multicenter [CONFIRM] Registry). Am J Cardiol. 2019 May 1;123(9):1435-1442. doi: 10.1016/j.amjcard.2019.01.055. Epub 2019 Feb 10. PMID 30850210
- [Background] Al'Aref SJ, Maliakal G, Singh G, van Rosendael AR, Ma X, Xu Z, Alawamlh OAH, Lee B, Pandey M, Achenbach S, Al-Mallah MH, Andreini D, Bax JJ, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJW, Cury RC, DeLago A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann PA, Kim YJ, Leipsic JA, Maffei E, Marques H, Goncalves PA, Pontone G, Raff GL, Rubinshtein R, Villines TC, Gransar H, Lu Y, Jones EC, Pena JM, Lin FY, Min JK, Shaw LJ. Machine learning of clinical variables and coronary artery calcium scoring for the prediction of obstructive coronary artery disease on coronary computed tomography angiography: analysis from the CONFIRM registry. Eur Heart J. 2020 Jan 14;41(3):359-367. doi: 10.1093/eurheartj/ehz565. PMID 31513271
- [Background] Han D, Beecy A, Anchouche K, Gransar H, Dunham PC, Lee JH, Achenbach S, Al-Mallah MH, Andreini D, Berman DS, Bax JJ, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJW, Cury RC, DeLago A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann PA, Kim YJ, Leipsic JA, Maffei E, Marques H, de Araujo Goncalves P, Pontone G, Raff GL, Rubinshtein R, Villines TC, Lu Y, Pena JM, Shaw LJ, Min JK, Lin FY. Risk Reclassification With Coronary Computed Tomography Angiography-Visualized Nonobstructive Coronary Artery Disease According to 2018 American College of Cardiology/American Heart Association Cholesterol Guidelines (from the Coronary Computed Tomography Angiography Evaluation for Clinical Outcomes : An International Multicenter Registry [CONFIRM]). Am J Cardiol. 2019 Nov 1;124(9):1397-1405. doi: 10.1016/j.amjcard.2019.07.045. Epub 2019 Aug 23. PMID 31547994
- [Background] Gnanenthiran SR, Naoum C, Leipsic JA, Achenbach S, Al-Mallah MH, Andreini D, Bax JJ, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJW, Cury RC, DeLago A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufman PA, Kim YJ, Maffei E, Marques H, de Araujo Goncalves P, Pontone G, Raff GL, Rubinshtein R, Shaw LJ, Villines TC, Gransar H, Lu Y, Jones EC, Pena JM, Lin FY, Kritharides L, Min JK. Long-term prognostic utility of computed tomography coronary angiography in older populations. Eur Heart J Cardiovasc Imaging. 2019 Nov 1;20(11):1279-1286. doi: 10.1093/ehjci/jez067. PMID 30993334
- [Background] Schulman-Marcus J, Lin FY, Gransar H, Berman D, Callister T, DeLago A, Hadamitzky M, Hausleiter J, Al-Mallah M, Budoff M, Kaufmann P, Achenbach S, Raff G, Chinnaiyan K, Cademartiri F, Maffei E, Villines T, Kim YJ, Leipsic J, Feuchtner G, Rubinshtein R, Pontone G, Andreini D, Marques H, Chang HJ, Chow BJW, Cury RC, Dunning A, Shaw L, Min JK. Coronary revascularization vs. medical therapy following coronary-computed tomographic angiography in patients with low-, intermediate- and high-risk coronary artery disease: results from the CONFIRM long-term registry. Eur Heart J Cardiovasc Imaging. 2017 May 1;18(8):841-848. doi: 10.1093/ehjci/jew287. PMID 28329294
- [Background] Deseive S, Shaw LJ, Min JK, Achenbach S, Andreini D, Al-Mallah MH, Berman DS, Budoff MJ, Callister TQ, Cademartiri F, Chang HJ, Chinnaiyan K, Chow BJ, Cury RC, DeLago A, Dunning AM, Feuchtner G, Kaufmann PA, Kim YJ, Leipsic J, Marques H, Maffei E, Pontone G, Raff G, Rubinshtein R, Villines TC, Hausleiter J, Hadamitzky M. Improved 5-year prediction of all-cause mortality by coronary CT angiography applying the CONFIRM score. Eur Heart J Cardiovasc Imaging. 2017 Mar 1;18(3):286-293. doi: 10.1093/ehjci/jew195. PMID 28363203
- [Derived] Gebhard C, Maredziak M, Messerli M, Buechel RR, Lin F, Gransar H, Achenbach S, Al-Mallah MH, Andreini D, Bax JJ, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJW, Cury RC, DeLago A, Feuchtner G, Hadamitzky M, Hausleiter J, Kim YJ, Leipsic J, Maffei E, Marques H, Goncalves PA, Pontone G, Raff GL, Rubinshtein R, Shaw LJ, Villines TC, Lu Y, Jones EC, Pena JM, Min JK, Kaufmann PA. Increased long-term mortality in women with high left ventricular ejection fraction: data from the CONFIRM (COronary CT Angiography EvaluatioN For Clinical Outcomes: An InteRnational Multicenter) long-term registry. Eur Heart J Cardiovasc Imaging. 2020 Apr 1;21(4):363-374. doi: 10.1093/ehjci/jez321. PMID 31985803
- [Derived] Opolski MP, Gransar H, Lu Y, Achenbach S, Al-Mallah MH, Andreini D, Bax JJ, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJ, Cury RC, DeLago A, Feuchtner GM, Hadamitzky M, Hausleiter J, Kaufmann PA, Kim YJ, Leipsic JA, Maffei EC, Marques H, Pontone G, Raff G, Rubinshtein R, Shaw LJ, Villines TC, Gomez M, Jones EC, Pena JM, Min JK, Lin FY. Prognostic value of chronic total occlusions detected on coronary computed tomographic angiography. Heart. 2019 Feb;105(3):196-203. doi: 10.1136/heartjnl-2017-312907. Epub 2018 Jul 30. PMID 30061160
- [Derived] Naoum C, Berman DS, Ahmadi A, Blanke P, Gransar H, Narula J, Shaw LJ, Kritharides L, Achenbach S, Al-Mallah MH, Andreini D, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow B, Cury RC, DeLago A, Dunning A, Feuchtner G, Hadamitzky M, Hausleiter J, Kaufmann PA, Kim YJ, Maffei E, Marquez H, Pontone G, Raff G, Rubinshtein R, Villines TC, Min J, Leipsic J. Predictive Value of Age- and Sex-Specific Nomograms of Global Plaque Burden on Coronary Computed Tomography Angiography for Major Cardiac Events. Circ Cardiovasc Imaging. 2017 Mar;10(3):e004896. doi: 10.1161/CIRCIMAGING.116.004896. PMID 28292858
- [Derived] Opolski MP, O Hartaigh B, Berman DS, Budoff MJ, Achenbach S, Al-Mallah M, Andreini D, Cademartiri F, Chang HJ, Chinnaiyan K, Chow BJ, Hadamitzky M, Hausleiter J, Feuchtner G, Kim YJ, Kaufmann PA, Leipsic J, Maffei E, Pontone G, Raff G, Shaw LJ, Villines TC, Min JK. Current trends in patients with chronic total occlusions undergoing coronary CT angiography. Heart. 2015 Aug;101(15):1212-8. doi: 10.1136/heartjnl-2014-306616. Epub 2015 Jun 15. PMID 26076936
- [Derived] Chow BJ, Small G, Yam Y, Chen L, McPherson R, Achenbach S, Al-Mallah M, Berman DS, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Cheng VY, Chinnaiyan K, Cury R, Delago A, Dunning A, Feuchtner G, Hadamitzky M, Hausleiter J, Karlsberg RP, Kaufmann PA, Kim YJ, Leipsic J, LaBounty T, Lin F, Maffei E, Raff GL, Shaw LJ, Villines TC, Min JK; CONFIRM Investigators. Prognostic and therapeutic implications of statin and aspirin therapy in individuals with nonobstructive coronary artery disease: results from the CONFIRM (COronary CT Angiography EvaluatioN For Clinical Outcomes: An InteRnational Multicenter registry) registry. Arterioscler Thromb Vasc Biol. 2015 Apr;35(4):981-9. doi: 10.1161/ATVBAHA.114.304351. Epub 2015 Feb 12. PMID 25676000